CLINICAL TRIAL: NCT05584475
Title: Mindful Awareness Practices for ADHD (MAPs): Pilot Open Trial
Brief Title: Mindful Awareness Practices for ADHD Pilot Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0399
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Treatment (Experimental): This arm consists of the mindfulness treatment that will be administered to all participants in the single-arm open trial.
  Interventions: Behavioral: Mindful Awareness Practices (MAPs)

INTERVENTIONS:
Behavioral: Mindful Awareness Practices (MAPs) — MAPs is an 8-session, group-based approach for individuals with ADHD to improve attentional difficulties and related impairments by enhancing attending to and accepting experiences in the present moment. Sessions typically last between 60 and 90 minutes, though may last up to 120 minutes.

SUMMARY:
It is estimated that 25-40% of youth with ADHD have co-occurring cognitive disengagement syndrome (CDS; previously sluggish cognitive tempo), a set of behavioral symptoms characterized by excessive daydreaming, slowed thinking, and mental confusion and fogginess. A growing body of research demonstrates CDS to be associated with functional impairment above and beyond that which can be accounted for by ADHD severity. However, no treatment currently exists that directly targets CDS symptoms. This is a critical clinical and scientific gap, leaving youth with ADHD and co-occurring CDS at risk for experiencing negative immediate and long-term outcomes. In considering intervention approaches, mindfulness meditation involves regular practice to catch oneself when the mind wanders, and may thus an ideal intervention for youth with CDS. However, mindfulness interventions, including the Mindful Awareness Practices (MAPs) for ADHD, have never been tested in adolescents with ADHD and co-occurring CDS specifically. This study will recruit up to 15 adolescents with ADHD and co-occurring CDS symptoms to enroll in an open trial of MAPs to evaluate its feasibility, acceptability, and preliminary efficacy. Findings will provide key pilot data regarding treatment of CDS in adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Between 13 and 17 years of age at the first MAPs session.
2. Estimated IQ ≥ 80 as assessed by the Kaufman Brief Intelligence Test, Second Edition (KBIT-2).
3. Meet full DSM-5 criteria for ADHD (per protocol).
4. SCT Total score >85th percentile (T-score >60) on the Child and Adolescent Behavior Inventory (CABI) SCT Module.
5. Sufficient English language ability necessary to complete study measures and intervention per parent and/or research staff judgment.
6. If applicable: If the adolescent is taking a medication for ADHD or another psychiatric disorder (e.g., anxiety, depression), the adolescent must be on a stable medication dose/schedule for at least one month, and families will also be asked to not change/add medications the adolescent takes during the intervention period.

Exclusion Criteria:

1. Children who have participated in behavioral therapy treatment in the past year will be ineligible.
2. Children with a parent-report diagnosis of autism spectrum disorder, bipolar disorder, obsessive-compulsive disorder, or psychosis will be excluded.
3. Significant visual, hearing, or speech impairment not helped with corrective or assistive devices (e.g., glasses, hearing aids) per parent report or study staff judgment.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change in mindfulness: Child and Adolescent Mindfulness Measure (CAMM) | Immediately after the intervention
  Mindfulness measured using the adolescent-completed Child and Adolescent Mindfulness Measure (CAMM). Scores range from 0 to 40 (higher = worse).

SECONDARY OUTCOMES:
Change in mind wandering: Mind-Wandering Questionnaire (MWQ) | Immediately after the intervention
  Mind wandering measured using the adolescent-completed Mind-Wandering Questionnaire (MWQ). SCores range from 5 to 30 (higher = worse).
Change in cognitive disengagement syndrome (CDS) symptoms: Child Concentration Inventory, Second Edition (CCI-2) | Immediately after the intervention
  CDS symptoms measured using the adolescent-completed Child Concentration Inventory, Second Edition (CCI-2). Scores range from 0 to 48 (higher = worse).
Change in attention-deficit/hyperactivity disorder (ADHD) symptoms: Vanderbilt ADHD Diagnostic Rating Scale (VADRS) | Immediately after the intervention
  ADHD symptoms measured using the parent-completed Vanderbilt ADHD Diagnostic Rating Scale (VADRS). Scores range from 0 to 27 (higher = worse).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Becker, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States